CLINICAL TRIAL: NCT06575582
Title: Digital Navigators for Acceptance and Competence Development with Mental Health Apps
Acronym: DigiNavi
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medizinische Hochschule Brandenburg Theodor Fontane (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other); Hannover Medical School (Other)
Responsible Party: Principal Investigator, Laura Uchtmann, M.Sc. Laura Uchtmann, Medizinische Hochschule Brandenburg Theodor Fontane
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 00034327
Record Dates: First submitted 2024-08-22; First posted 2024-08-28 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Acceptability of Health Care; Engagement, Patient; Nurse's Role; Mental Disorder
Keywords: digital health; ehealth; mhealth; mental health; health literacy
MeSH Terms: conditions — Patient Acceptance of Health Care; Patient Participation; Mental Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The use of digital navigators in multi-professional treatment teams is a complex intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Exploratory preliminary study (No Intervention): General practitioners (n = 10), outpatient psychiatrists and psychologists (n = 10) and their patients (n = 20) will be involved. First, partly structured interviews will be conducted with the general practitioners and the psychiatric/psychological professionals as well as the patients they treat in order to record their perspectives on digital health services and the role of digital navigators. In parallel, focus groups will be organized with all three main groups to understand their opinions, concerns and expectations regarding the use of digital health applications and digital navigators. The data collection for the preliminary study extends over a period of 3 months (October - December 2024).
- Training (Experimental): Staff members (n = 6) of participating study cites will be trained to become Digital Navigators. The recruitment and training of the digital navigators will take place over a period of 4 months (October 2024 to January 2025).
  Interventions: Behavioral: Training for Digital Navigators
- Treatment team and patient support (Experimental): The Digital Navigators support the treatment teams in the study centers in the selection and integration of suitable apps and digital health applications (DiGAs). The selected patients (n = 48, 8 per center) are accompanied and supported by the trained navigators for 12 weeks to find a suitable app for them and integrate it into their treatment. A total period of 3 months is planned for both the recruitment of patients and the implementation off the intervention (December 2024 to February 2025).
  Interventions: Behavioral: Support from Digital Navigators to Treatment Team; Behavioral: Support from Digital Navigators to Patients

INTERVENTIONS:
Behavioral: Support from Digital Navigators to Treatment Team — The trained professionals (the Digital Navigators) support the treatment teams in the study centers in the selection and integration of suitable apps and digital health applications (DiGAs).
  Arms: Treatment team and patient support
Behavioral: Support from Digital Navigators to Patients — The trained professionals (the Digital Navigators) accompany and support the selected patients to find a suitable app for them and integrate it into their treatment.
  Arms: Treatment team and patient support
Behavioral: Training for Digital Navigators — The training takes place in the six study centers and is preferably aimed at medical assistants.
  Arms: Training

SUMMARY:
The goal of this clinical trial is to learn if and how so called "Digital Navigators" (DN) can help general practitioners, outpatient psychiatrists and psychologists as well as their treated patients to use digital mental health apps (DiGAs) and integrate it into their treatment. The main questions it aims to answer are:

* What are the chances and implementation barriers of DN?
* What are the acceptance and expectations towards DN?
* Do DN affect the psychological health of patients?
* Do DN affect the digital health literacy and technical competence of participants?

Employees of medical teams (e.g. medical assistants) receive training to become a DN. Afterwards patients are accompanied and supported by the DN for 12 weeks to select and use a suitable app for their mental disorder.

DETAILED DESCRIPTION:
The study aims to promote the use of digital health applications (DiGAs) to improve mental health and provide timely treatment for underserved populations. Currently, DiGAs are only used by a small proportion of patients and practitioners in Germany. In order to solve this care problem, employees of medical teams, such as medical assistants, are to be trained as so-called 'digital navigators'. These digital navigators support stakeholders in the selection and use of mental health apps, impart the necessary digital skills, improve adherence and relieve the burden on those providing treatment.

As part of the pilot project, digital navigators will be implemented as an example in GP and outpatient psychiatric care in a rural region of Brandenburg. Firstly, a preliminary study will be conducted to determine the acceptance and expectations of the digital navigators using interviews and focus groups. The researchers then complete a training program at Harvard Medical School and adapt the 'Harvard Digital Navigator Training' to the German framework conditions. This adaptation process is supported by discussion groups with patients and practitioners.

In the next step, medical assistants in six study centres will receive the adapted training. A central tool available to them is the DiGAnavigator.de website, a guide for DiGAs. The digital navigators help with the integration of DiGAs into the treatment of 48 patients with mental illnesses and accompany them over a period of 12 weeks.

Finally, the implementation will be evaluated. The evaluation analyses the implementation hurdles and the effects on the eHealth literacy of patients and professionals. The eHealth Literacy Scale (eHeals) and the Digital Health Literacy Index (DHLI) will be used for this purpose. An accompanying process evaluation analyses the acceptance, effects and implementation barriers of the digital navigators. In addition, both patients and staff are surveyed regarding their digital and technical skills as well as their willingness and ability to change before and after the intervention. Furthermore, the severity of the patients' illness will be recorded and compared before and after the intervention using validated scales. To ensure sustainable implementation, the long-term aim is to provide accredited training to become a digital navigator.

ELIGIBILITY:
Inclusion Criteria:

* Main diagnosis according to ICD 10 F00-F69, F80-F99
* Capacity to consent is given
* Sufficient language skills for an interview in German
* Participants have access to modern digital hardware (smartphone)
* Basic knowledge of how to operate a smartphone

Exclusion Criteria:

* Acute danger to self or others
* Patients have received prompt (<= 3 weeks) qualified psychiatric or psychotherapeutic treatment
* Severe organic brain diseases with cognitive deficits
* Intellectual disability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-07-14 (Estimated)

PRIMARY OUTCOMES:
Digital health literacy (focus: digital information retrieval skills) | Before (T0) and after completion of the 12-week intervention (T1)
  Using the self-report rating inventory eHealth Literacy Scale (eHeals). Total score ranges from 8 to 40, with higher scores representing higher self-perceived eHealth literacy.
Digital health literacy (focus: digital interactive skills) | Before (T0) and after completion of the 12-week intervention (T1)
  Using a performance-based rating inventory Digital Health Literacy Index (DHLI). Total score ranges from 0 to 7, with higher scores representing a greater ability to operate digital devices and read and write in web-based modes.
Acceptance towards Digital Navigators | Before the intervention (T0)
  Qualitative questions using semi-structured interviews
Expectations towards Digital Navigators | Before the intervention (T0)
  Qualitative questions using focus groups
Expectations towards Digital Navigators | Before the intervention (T0)
  Qualitative questions using semi-structured interviews
Acceptance towards Digital Navigators | Before the intervention (T0)
  Qualitative questions using focus groups

SECONDARY OUTCOMES:
Willingness and competence to change | Before (T0) and after completion of the 12-week intervention (T1)
  Using the self-report rating inventory "Readiness for Change". Total score ranges from 0 to 172, with higher scores representing higher self-perceived willingness and competence to change.
Digital competence | Before (T0) and after completion of the 12-week intervention (T1)
  Using the self-report rating inventory ICT Self-Concept Scale. Total score ranges from 25 to 150, with higher scores representing higher self-perceived digital competence.
Technical competence | Before (T0) and after completion of the 12-week intervention (T1)
  Using the self-report rating inventory "Kurzskala Technikbereitschaft" (TB, technology commitment). Total score ranges from 12 to 60, with higher scores representing higher self-perceived technical competence.
Psychological Health of Patients (level of functioning) | After completion of the 12-week intervention (T1)
  Using the self-report rating inventory Global Assessment of Functioning (GAF). Total score ranging from 0-100, with a higher score indicating a higher level of functioning.
Psychological Health of Patients (symptom severity, treatment response and the efficacy of treatment) | Before (T0) and after completion of the 12-week intervention (T1)
  Using the self-report rating inventory Clinical Global Impression (CGI); Measuring three dimensions: severity of illness (score 1-7, with a higher score indicating a more severe illness), global improvement (score 1-7, with a higher score indicating a worsening of symptoms) and efficacy (measured with 4×4 rating scale (ranging from 01 - 16) that assesses the therapeutic effect of treatment and associated side effects; e.g. 01 = no side effects; vast improvement; 16 = severe side effects; unchanged or worse condition)
Psychological Health of Patients (depressive symptoms; self-report) | Before (T0) and after completion of the 12-week intervention (T1)
  Using the self-report rating inventory Beck's Depression Inventory (BDI); Total score 0-63, with higher scores representing more severe depressive symptoms.
Psychological Health of Patients (depressive symptoms; clinician-administered) | Before (T0) and after completion of the 12-week intervention (T1)
  Using the clinician-administered rating inventory Hamilton Depression Scale (HAMD); Total score 0-52, with higher scores representing more severe depressive symptoms.
Psychological Health of Patients (anxiety) | Before (T0) and after completion of the 12-week intervention (T1)
  Using the clinician-administered rating inventory Hamilton Anxiety Scale (HAMA); Total score 0-56, with higher scores representing more severe anxiety symptoms.
Psychological Health of Patients (insomnia) | Before (T0) and after completion of the 12-week intervention (T1)
  Using the self-report rating inventory Insomnia Severity Index (ISI); Total score 0-28, with higher scores representing more severe insomia symptoms.
Identification of implementation barriers to the introduction of digital navigators | After completion of the 12-week intervention (T1)
  Qualitative questions using semi-structured interviews
Identification of implementation barriers to the introduction of digital navigators | After completion of the 12-week intervention (T1)
  Qualitative questions using focus groups
Use of Digital Health Applications and the effects of counseling and support by Digital Navigators | After completion of the 12-week intervention (T1)
  Qualitative questions using semi-structured interviews
Use of Digital Health Applications and the effects of counseling and support by Digital Navigators | After completion of the 12-week intervention (T1)
  Qualitative questions using focus groups

CONTACTS AND LOCATIONS:
Overall Officials: Martin Heinze, Prof, Study Chair — Medizinische Hochschule Brandenburg Theodor Fontane
Locations (6):
- Germany (6):
  - Praxis Brandenburg an der Havel, Brandenburg, Brandenburg
  - Praxis Eberswalde, Eberswalde, Brandenburg
  - Psychiatrische Institutsambulanz (PIA) Fürstenwalde, Fürstenwalde, Brandenburg
  - Praxis Fürstenwalde, Fürstenwalde, Brandenburg
  - Psychiatrische Institutsambulanz (PIA) Rüdersdorf, Rüdersdorf, Brandenburg
  - Psychiatrische Institutsambulanz (PIA) Strausberg, Strausberg, Brandenburg

IPD SHARING:
Plan to Share IPD: No
We have decided not to make the individual participant data (IPD) publicly available in order to ensure the highest level of data protection and confidentiality. Although all data will be properly anonymized, we want to ensure that no conclusions can be drawn about individual participants, not even indirectly. The protection of study participants' personal data is a top priority for us. Therefore, for ethical and data protection reasons, it is more responsible not to make the IPD publicly accessible.

REFERENCES:
- [Derived] Schwarz J, Chen K, Dashti H, Heinze M, Schonbeck J, Schubert D, Senst B, Speck J, Torous J, Wolff J, Uchtmann L, Meier-Diedrich E. Piloting Digital Navigators to Promote Acceptance and Engagement With Digital Mental Health Apps in German Outpatient Care: Protocol for a Multicenter, Single-Group, Observational, Mixed Methods Interventional Study (DigiNavi). JMIR Res Protoc. 2025 Sep 25;14:e67655. doi: 10.2196/67655. PMID 40996088
- See also: Information about study from German Federal Ministry of Health (in German) — https://www.bundesgesundheitsministerium.de/ministerium/ressortforschung/handlungsfelder/forschungsschwerpunkte/pilotvorhaben-zur-implementierung-und-verstetigung-von-digital-health-ansaetzen/diginavi.html
- See also: Official DigiNavi Website — https://www.diginavi.de/en/